CLINICAL TRIAL: NCT06737458
Title: Serratus Anterior Plane Block Versus Erector Spinae Plane Block With Dexmedetomidine Added to Bupivacaine for Ultrasound-Guided Pain Management After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hend Saad Rizk Farhat, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelshiekh University, Kafrelshiekh, Egypt, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-438
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Serratus Anterior Plane Block; Erector Spinae Plane Block; Dexmedetomidine; Bupivacaine; Ultrasound; Pain Management; Mastectomy
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus anterior plane block group (Active Comparator): Patients received serratus anterior plane block on the operated side with bupivacaine 0.25% plus 0.5 µg/kg dexmedetomidine in 30 ml.
  Interventions: Drug: Bupivacaine + Dexmedetomidine
- Erector spinae plane block group (Experimental): Patients received erector spinae plane block at T5 on the operated side and will receive bupivacaine 0.25% plus 0.5 µg/kg dexmedetomidine in 30 ml.
  Interventions: Drug: Bupivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine + Dexmedetomidine — Patients received serratus anterior plane block on the operated side with bupivacaine 0.25% plus 0.5 µg/kg dexmedetomidine in 30 ml.
  Other Names: Serratus anterior plane block
  Arms: Serratus anterior plane block group
Drug: Bupivacaine + Dexmedetomidine — Patients received erector spinae plane block at T5 on the operated side and will receive bupivacaine 0.25% plus 0.5 µg/kg dexmedetomidine in 30 ml.
  Other Names: Erector spinae plane block
  Arms: Erector spinae plane block group

SUMMARY:
This study aimed to compare the serratus plane block versus the erector spinae plane block with dexmedetomidine added to bupivacaine for acute pain management after breast surgeries.

DETAILED DESCRIPTION:
Approximately 40-60% of breast surgery patients endure severe acute postoperative pain, with over 10% of patients experiencing severe pain for six to twelve months (post-mastectomy pain syndrome).

Dexmedetomidine has analgesic properties, which could be related to the stimulation of α2 adrenoceptors, inhibition of nerve conduction through C and Aδ fibers, and the local release of encephalin.

Serratus plane block (SPB) is an effective approach for breast surgery analgesia due to its simplicity of delivery, minimal risk of adverse effects, and ability to provide significant pain relief.

The erector spinae plane block (ESPB) is one of the emerging regional techniques for managing postoperative pain. ESPB can be given unilaterally during modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >20 years.
* Patient's approval.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Patients underwent breast surgeries.

Exclusion Criteria:

* Known allergy to local anesthetics, opioids, or dexmedetomidine medications.
* Advanced heart block, ventricular dysfunction.
* Skin infection at the site of injection.
* Pre-existing chronic pain.
* Coagulopathies, significant liver or renal insufficiency.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients underwent breast surgeries.
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Total dose of pethidine consumption | 24 hours postoperatively
  Patients get 1 g paracetamol IV like clockwork. Salvage absence of pain as bolus IV pethidine at 0.5 mg/kg was managed if NRS > 3

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  In case the cruel blood vessel weight (Outline) or heart rate (HR) went over 20% of pattern values, additional bolus dosages of 0.5 µg/kg IV fentanyl were given.
Heart rate | Every 15 minutes until the end of the surgery (Up to 2 hours)
  Heart rate was measured preoperatively and intraoperatively every 15 minutes until the end of the surgery.
Mean arterial pressure | Every 15 minutes until the end of the surgery (Up to 2 hours)
  Mean arterial pressure was measured preoperatively and intraoperatively every 15 minutes until the end of the surgery.
Degree of pain | 24 hours postoperatively
  Each patient was instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS was assessed at post anesthesia care unit, 1, 2, 6, 12, 18, and 24 hours postoperatively
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as hypotension, bradycardia, and postoperative nausea and vomiting (PONV) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.